CLINICAL TRIAL: NCT04789161
Title: Comparison of Double-kissing Crush and Double-kissing Culotte Stenting in Patients With True Bifurcation Lesion
Brief Title: Comparison of Double-kissing Crush and Double-kissing Culotte Stenting
Status: Completed | Type: Observational
Sponsor: Istanbul Mehmet Akif Ersoy Educational and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Serkan Kahraman, Associate Professor, Istanbul Mehmet Akif Ersoy Educational and Training Hospital
Other Study IDs: IMAEETH-2
Record Dates: First submitted 2021-03-05; First posted 2021-03-09 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- double kissing crush stenting: patients with true bifurcation lesion undergoing double kissing crush stenting
  Interventions: Procedure: double kissing crush stenting
- double kissing culotte stenting: patients with true bifurcation lesion undergoing double kissing culotte stenting
  Interventions: Procedure: double kissing culotte stenting

INTERVENTIONS:
Procedure: double kissing crush stenting — Patients with true bifurcation lesion treating with double kissing crsuh stenting technique
  Groups: double kissing crush stenting
Procedure: double kissing culotte stenting — Patients with true bifurcation lesion treating with double kissing culotte stenting technique
  Groups: double kissing culotte stenting

SUMMARY:
True bifurcation lesions (TBLs) are not rare clinical conditions and may be associated with adverse cardiovascular outcomes due to their complex anatomy and the variety of interventional therapy. Although the provisional stenting is still effective in suitable lesions, double stent techniques can be required in selected patients. In previous studies, double kissing crush (DK-crush) stenting was revealed as superior to provisional stenting in TBL of left main coronary artery. Additionally, in recent studies, double kissing approach facilitates and highlights double kissing culotte (DK-culotte) stenting with lower stent malapposition compared to DK-crush stenting. However, to the best of our knowledge, there is no study about comparing DK-crush and DK-culotte stenting in TBLs. Our aim in this study is to compare DK-crush and DK-culotte stenting in patients with TBL.

ELIGIBILITY:
Inclusion Criteria:

* Patients with de novo true bifurcation lesion (Medina classification 1,1,1 or 0,1,1 or 1,0,1)
* The main vessel diameter is least 2.5 mm and the side branch diameter is at least 2.25 mm

Exclusion Criteria:

* Patients presenting with ST segment elevation myocardial infarction, cardiogenic shock and Killip class III-IV heart failure
* Patients with a history of coronary artery bypass grafting surgery
* Patients with a chronic total occlusion in the bifurcation area
* Lesions with severe calcification that needs additional intervention such as atherectomy
* Patients who are not suitable to use long term dual antiplatelet therapy and patients not participating in clinical follow-up
* Patients with hematological disorders, malignancy, end stage renal (GFR<30 ml/min) and hepatic failure
* Patients with active bleeding
* Pregnant women
* Patients with life-expectancy < 1 year

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stable or unstable angina pectoris or patients with non-ST segment elevation myocardial infarction undergoing percutaneous coronary intervention and performing double stent techniques (DK-crush or DK-culotte) are included in this study.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-05-04 (Actual)

PRIMARY OUTCOMES:
MACE (major adverse cardiovascular events) | 12 months
  target vessel revascularization, myocardial infarction and cardiac death

SECONDARY OUTCOMES:
MACCEs (major adverse cerebral and cardiovascular events) | 12, 24, 36 months
  all cause death, myocardial infarction, target lesion revascularization, target lesion revascularization, in-stent thrombosis and/or restenosis, stroke
target lesion failure | 24, 36 months
  myocardial infarction, cardiac death

OTHER OUTCOMES:
contrast induced nephropathy | 12 months
  25 percent (%) increase in serum creatinine level from baseline or a 0.5 mg/dL increase in absolute serum creatinine value within 72 hours after percutaneous coronary intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Mehmet Akif Ersoy Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Steigen TK, Maeng M, Wiseth R, Erglis A, Kumsars I, Narbute I, Gunnes P, Mannsverk J, Meyerdierks O, Rotevatn S, Niemela M, Kervinen K, Jensen JS, Galloe A, Nikus K, Vikman S, Ravkilde J, James S, Aaroe J, Ylitalo A, Helqvist S, Sjogren I, Thayssen P, Virtanen K, Puhakka M, Airaksinen J, Lassen JF, Thuesen L; Nordic PCI Study Group. Randomized study on simple versus complex stenting of coronary artery bifurcation lesions: the Nordic bifurcation study. Circulation. 2006 Oct 31;114(18):1955-61. doi: 10.1161/CIRCULATIONAHA.106.664920. Epub 2006 Oct 23. PMID 17060387
- [Result] Colombo A, Bramucci E, Sacca S, Violini R, Lettieri C, Zanini R, Sheiban I, Paloscia L, Grube E, Schofer J, Bolognese L, Orlandi M, Niccoli G, Latib A, Airoldi F. Randomized study of the crush technique versus provisional side-branch stenting in true coronary bifurcations: the CACTUS (Coronary Bifurcations: Application of the Crushing Technique Using Sirolimus-Eluting Stents) Study. Circulation. 2009 Jan 6;119(1):71-8. doi: 10.1161/CIRCULATIONAHA.108.808402. Epub 2008 Dec 22. PMID 19103990
- [Result] Hildick-Smith D, de Belder AJ, Cooter N, Curzen NP, Clayton TC, Oldroyd KG, Bennett L, Holmberg S, Cotton JM, Glennon PE, Thomas MR, Maccarthy PA, Baumbach A, Mulvihill NT, Henderson RA, Redwood SR, Starkey IR, Stables RH. Randomized trial of simple versus complex drug-eluting stenting for bifurcation lesions: the British Bifurcation Coronary Study: old, new, and evolving strategies. Circulation. 2010 Mar 16;121(10):1235-43. doi: 10.1161/CIRCULATIONAHA.109.888297. Epub 2010 Mar 1. PMID 20194880
- [Result] Chen SL, Zhang JJ, Han Y, Kan J, Chen L, Qiu C, Jiang T, Tao L, Zeng H, Li L, Xia Y, Gao C, Santoso T, Paiboon C, Wang Y, Kwan TW, Ye F, Tian N, Liu Z, Lin S, Lu C, Wen S, Hong L, Zhang Q, Sheiban I, Xu Y, Wang L, Rab TS, Li Z, Cheng G, Cui L, Leon MB, Stone GW. Double Kissing Crush Versus Provisional Stenting for Left Main Distal Bifurcation Lesions: DKCRUSH-V Randomized Trial. J Am Coll Cardiol. 2017 Nov 28;70(21):2605-2617. doi: 10.1016/j.jacc.2017.09.1066. Epub 2017 Oct 30. PMID 29096915
- [Result] Toth GG, Sasi V, Franco D, Prassl AJ, Di Serafino L, Ng JCK, Szanto G, Schneller L, Ang HY, Plank G, Wijns W, Barbato E. Double-kissing culotte technique for coronary bifurcation stenting. EuroIntervention. 2020 Oct 9;16(9):e724-e733. doi: 10.4244/EIJ-D-20-00130. PMID 32338608
- [Derived] Kahraman S, Cizgici AY, Guner A, Tasbulak O, Panc C, Dogan AC, Ulutas AE, Gurbak I, Bulut U, Avci Y, Demir AR, Yalcin AA, Kalkan AK, Erturk M. Clinical Outcomes of Double-Kissing Crush or Double-Kissing Culotte in Nonleft Main Bifurcation Lesions: The ROUTE Trial. Circ Cardiovasc Interv. 2024 Nov;17(11):e014616. doi: 10.1161/CIRCINTERVENTIONS.124.014616. Epub 2024 Oct 24. PMID 39445416